CLINICAL TRIAL: NCT03691090
Title: PD-1 Antibody SHR-1210 Combined With Paclitaxel and Cisplatin Versus Placebo Combined With Paclitaxel and Cisplatin as First-line Therapy for Advanced Esophageal Cancer: a Randomized, Double-blinded, Controlled, Multi-center Phase III Trial
Brief Title: Study of SHR-1210 in Combination With Chemotherapy in Advanced Esophageal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1210-III-306
Record Dates: First submitted 2018-09-21; First posted 2018-10-01 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-06

CONDITIONS: Advanced Esophageal Cancer
Keywords: PD-1Antibody; advanced esophageal cancer; paclitaxel; cisplatin
MeSH Terms: interventions — camrelizumab; Paclitaxel; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-1210 + paclitaxel + cisplatin (Experimental): Paclitaxel 175mg/m2, Day 1，cisplatin 75mg/m2，Day 1，SHR-1210 200mg，Day 2，every 3 weeks, maximum 6 cycles, then SHR-1210 maintenance
  Interventions: Drug: SHR-1210; Drug: paclitaxel; Drug: cisplatin
- placebo+paclitaxel + cisplatin (Active Comparator): Paclitaxel 175mg/m2, Day 1，cisplatin 75mg/m2，Day 1，placebo，Day 2，every 3 weeks, maximum 6 cycles, then placebo maintenance
  Interventions: Drug: Placebo; Drug: paclitaxel; Drug: cisplatin

INTERVENTIONS:
Drug: SHR-1210 — SHR-1210 200mg
  Other Names: camrelizumab
  Arms: SHR-1210 + paclitaxel + cisplatin
Drug: Placebo — Placebo
  Arms: placebo+paclitaxel + cisplatin
Drug: paclitaxel — paclitaxel 175mg/m2
Drug: cisplatin — cisplatin 75mg/m2

SUMMARY:
This is a randomised, double-blinded, placebo-controlled, multi-center phase III trial, comparing the efficacy and safety of SHR-1210 + paclitaxel + cisplatin vs placebo+paclitaxel +cisplatin as 1L therapy for advanced esophageal cancer patients in China. SHR-1210 is a humanized anti-PD1 IgG4 monoclonal antibody.

DETAILED DESCRIPTION:
In this study, eligible subjects will be randomized into study arm or control arm. Treatment cycles of chemotherapy will be at most 6 cycles which would be decided by the investigators. Progression-free survival (PFS) assessed by the Independent Review Committee (IRC) and overall survival (OS) will be the primary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed unresectable local advanced/recurrent or metastasis esophageal squamous cell carcinoma;
2. No previous systemic anti-tumor treatment;
3. Subjects must have at least one measurable tumor lesion per RECIST 1.1;
4. Tissue samples should be provided for biomarkers (such as PD-L1) analysis;
5. ECOG: 0-1;
6. Adequate organ and bone marrow function;

Exclusion Criteria:

1. Allergic to monoclonal antibodies, any SHR-1210 components, paclitaxel, cisplatin and other platinum drugs;
2. Prior therapy as follow:

   1. Anti-PD-1 or anti-PD-L1;
   2. Any experimental drugs within 4 weeks of the first dose of study medication;
   3. Received major operations or serious injuries within 4 weeks of the first dose of study medication;
   4. Received last dose of anticancer therapy (including chemotherapy, radiotherapy, targeted therapy, etc.) within 4 weeks of the first dose of study medication;
3. Not recovered to ≤CTCAE 1 from adverse events (except for hair loss) due to a previously anti-tumor treatment;
4. Subjects with any active autoimmune disease or history of autoimmune disease;
5. Pregnancy or breast feeding;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 596 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
PFS assessed by IRC | approximately 22 months
  based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)
OS | approximately 22 months
  OS is defined as the time from registration to death due to any cause, or censored at date last known alive. Measured by the method of Kaplan and Meier.

SECONDARY OUTCOMES:
PFS assessed by investigators | approximately 22 months
  based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)
6 and 9 month OS rate | approximately 6 and 9 months
  OS is defined as the time from registration to death due to any cause, or censored at date last known alive. Measured by the method of Kaplan and Meier.
ORR | approximately 22 months
  based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)
DCR | approximately 22 months
  based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)
DoR | approximately 22 months
  based on response evaluation criteria in solid tumors 1.1 (RECIST 1.1)
AE | approximately 22 months
  adverse events

OTHER OUTCOMES:
Antidrug Antibodies (ADAs) | approximately 22 months
  To evaluate the incidence of ADAs against SHR-1210

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Principal Investigator — Cancer Center of Sun-Yat Sen University (CCSYSU); Qing Yang, Study Director — Jiangsu HengRui Medicine Co., Ltd.
Locations (1):
- Cancer Center of Sun-Yat Sen University (CCSYSU), Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang Y, Li C, Du K, Pengkhun N, Huang Z, Gong M, Li Y, Liu X, Li L, Wang D, Wang C, Chen F, Li J. Comparative analysis of immune checkpoint inhibitors in first-line treatment of esophageal squamous cell carcinoma: a network meta-analysis. Immunotherapy. 2023 Jul;15(10):737-750. doi: 10.2217/imt-2022-0236. Epub 2023 May 4. PMID 37139963
- [Derived] Luo H, Lu J, Bai Y, Mao T, Wang J, Fan Q, Zhang Y, Zhao K, Chen Z, Gao S, Li J, Fu Z, Gu K, Liu Z, Wu L, Zhang X, Feng J, Niu Z, Ba Y, Zhang H, Liu Y, Zhang L, Min X, Huang J, Cheng Y, Wang D, Shen Y, Yang Q, Zou J, Xu RH; ESCORT-1st Investigators. Effect of Camrelizumab vs Placebo Added to Chemotherapy on Survival and Progression-Free Survival in Patients With Advanced or Metastatic Esophageal Squamous Cell Carcinoma: The ESCORT-1st Randomized Clinical Trial. JAMA. 2021 Sep 14;326(10):916-925. doi: 10.1001/jama.2021.12836. PMID 34519801